CLINICAL TRIAL: NCT05188053
Title: Periarticular Bupivacaine + Meloxicam ER Solution Versus Standard Practice During Total Knee Arthroplasty: A Single Institution, Single-blinded, Randomized Clinical Trial
Brief Title: Periarticular Bupivacaine + Meloxicam ER Solution Versus Standard Practice During Total Knee Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Matthew P. Abdel, M.D., Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21-010044
Record Dates: First submitted 2021-12-27; First posted 2022-01-12 (Actual); Results first posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Total Knee Arthroplasty
MeSH Terms: interventions — bupivacaine-meloxicam drug combination; Ropivacaine; Epinephrine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- HTX-011 Treatment Group (Experimental): Subjects undergoing a total knee arthroplasty will receive HTX-011 (Zynrelef) for perioperative analgesia
  Interventions: Drug: HTX-011
- Standard Block Control Group (Active Comparator): Subjects undergoing a total knee arthroplasty will receive standard of care arthroplasty block for perioperative analgesia
  Interventions: Drug: ropivacaine , epinephrine , ketorolac diluted in sodium chloride

INTERVENTIONS:
Drug: HTX-011 — Single dose administration periarticular 400mg bupivacaine and 12mg meloxicam extended release solution
  Other Names: Zynrelef
  Arms: HTX-011 Treatment Group
Drug: ropivacaine , epinephrine , ketorolac diluted in sodium chloride — Single dose administration in 100cc of standard formulation, there is 225mg of ropivacaine 5mg/mL, 0.6mg epinephrine 1mg/mL, 30mg ketorolac 30mg/mL diluted in sodium chloride
  Other Names: Mayo Clinic standard arthroplasty block
  Arms: Standard Block Control Group

SUMMARY:
The purpose of this study is to compare an FDA-approved medication for post-operative pain control (HTX-011) to the standard of care institutional practice for periarticular analgesia after primary total knee arthroplasty (weight based dosing of Ropivacaine, epinephrine and ketorolac diluted with saline). We are doing this research study to find out if this new medication provides superior pain control within 72 hours following surgery.

ELIGIBILITY:
Inclusion Criteria:

* ASA classification I to III, older than or equal to 18 years old.
* Presenting for primary total knee replacement for degenerative joint disease.
* Patient capable of providing their own informed consent.

Exclusion Criteria:

* Vulnerable study populations including prisoners.
* Patients with a contralateral total knee arthroplasty < 2 years prior to the index procedure.
* Compromised health barring them from proceeding with surgery including acute or chronic kidney injury identified pre-operative.
* Patients unable to provide their own informed consent.
* Pregnancy.
* Patients with documented chronic pain syndromes.
* Patients with a history of prolonged daily opioids (more than 1 month) with an oral morphine equivalent of greater than 5mg/day.
* BMI > 45 kg/m^2.
* Allergies to any component of the study medications, including specific history of type 1 hypersensitivities to any NSAID.
* Patients with impaired cognitive function.
* Major systemic illnesses such as severe renal (estimated glomerular filtration rate less than 50ml/min), coronary artery disease requiring a bypass graft (CABG), other cardiac problems including congestive heart failure (CHF New York Heart Association class III to IV), or severe hepatic disorders defined as current or past diagnosis of acute/subacute liver necrosis, acute hepatic failure, chronic liver disease, liver abscess, hepatic coma, hepatorenal syndrome and other disorders of the liver.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 209 (Actual)
Dates: Start 2022-03-11 (Actual); Primary Completion 2024-04-18 (Actual); Study Completion 2024-04-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew P Abdel, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment for this study ran from 3/11/2022 until 4/9/2024 when the final patient was enrolled. Patients were enrolled from the Orthopedic clinical practice at Mayo Clinic.
Pre-assignment Details: An initial pilot of 18 patients ran from 3/11/2022 to 8/30/2022 after which a protocol change caused these patients to be withdrawn and not assigned to a treatment arm in the final study count. One additional patient was withdrawn prior to randomization as allergy results returned which excluded participation.
Period: Overall Study
Arm/Group | HTX-011 Treatment Group | Standard Block Control Group
Started | 95 | 95
Completed | 53 | 48
Not Completed | 42 | 47
Not completed — Lost to Follow-up | 23 | 30
Not completed — Protocol Violation | 16 | 16
Not completed — Physician Decision | 3 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HTX-011 Treatment Group | Standard Block Control Group | Total
Number analyzed (Participants) | 95 | 95 | 190
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.6 (8.1) | 69.9 (8.6) | 69.7 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 54 | 108
  Male | 41 | 41 | 82
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Pain Control at 72 Hours Postoperatively
Description: Area Under the Curve (AUC) of the graph for mean Numerical Rated Score (NRS) for pain (0-10) over time (0-72 hours) / NRS AUC 0-72. Pain scores were collected by patient self-report 15 times over the 72 hours after surgery, and averaged amongst the patients for each study arm.
  Lower values represent better pain control based on lower mean 0-10 pain scores over the 72 hour period after surgery. The minimum value is 0, meaning patients reported 0 pain on a 0-10 scale at all 15 time points within 72 hours. The maximum value would be 720, meaning patients reported a 10 for pain on a 0-10 scale at all 15 time points within 72 hours.
Time Frame: 72-hours postoperatively after total knee arthroplasty
Measure: Mean (Standard Deviation); unit: score on a scale * hours
Arm/Group | HTX-011 Treatment Group | Standard Block Control Group
Number analyzed (Participants) | 53 | 48
score on a scale * hours | 334 (16) | 370 (21)
Statistical Analysis 1: Comparison: HTX-011 Treatment Group vs Standard Block Control Group; Two-sample t-test with unequal variance. The null hypothesis is that there was no statistically significant difference between the two treatment groups based on a standard alpha value of 0.05; Test type: Other — Sample size calculations were performed to estimate the number of subjects needed to detect a 30% difference in NRS pain AUC scores between the study groups. 30% reduction in pain was considered the minimal clinically important difference in pain control based off previous pain research. A 30% reduction in pain would correspond with a difference of approximately 136 in area under the curve of mean pain over time; p = 0.170, t-test, 2 sided — a priori threshold p <0.05; assuming unequal variance

2. Secondary Outcome: Pain Control at 48 Hours Postoperatively
Description: Area Under the Curve (AUC) of the graph for mean Numerical Rated Score (NRS) for pain (0-10) over time (0-48 hours) / NRS AUC 0-48. Pain scores were collected by patient self-report 11 times over the 48 hours after surgery, and averaged amongst the patients for each study arm.
  Lower values represent better pain control based on lower mean 0-10 pain scores over the 48 hour period after surgery. The minimum value is 0, meaning patients reported 0 pain on a 0-10 scale at all 11 time points within 48 hours. The maximum value would be 480, meaning patients reported a 10 for pain on a 0-10 scale at all 11 time points within 48 hours
Time Frame: 48-hours postoperative total knee arthroplasty
Measure: Mean (Standard Deviation); unit: score on a scale * hours
Arm/Group | HTX-011 Treatment Group | Standard Block Control Group
Number analyzed (Participants) | 53 | 48
score on a scale * hours | 237 (14) | 268 (13)

3. Secondary Outcome: Opioid Consumption 72 Hours Postoperatively
Description: Total postoperative opioid consumption standardized into morphine milligram equivalents (MMEs)
Time Frame: 72-hours postoperative total knee arthroplasty
Population: patient who returned a complete pain diary
Measure: Mean (Full Range); unit: MME
Arm/Group | HTX-011 Treatment Group | Standard Block Control Group
Number analyzed (Participants) | 53 | 48
MME | 85 [0 to 238] | 77 [0 to 163]

4. Secondary Outcome: Opioid Consumption 48 Hours Postoperatively
Description: Total postoperative opioid consumption standardized into morphine milligram equivalents (MMEs)
Time Frame: 48 hours postoperative total knee arthroplasty
Population: patients who returned a completed pain diary
Measure: Mean (Full Range); unit: MME
Arm/Group | HTX-011 Treatment Group | Standard Block Control Group
Number analyzed (Participants) | 53 | 48
MME | 67 [0 to 163] | 60 [0 to 182]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from patient consent until 72 hours postoperatively.
Arm/Group | HTX-011 Treatment Group | Standard Block Control Group
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/48
Other Adverse Events (participants affected / at risk) | 1/53 | 2/48
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HTX-011 Treatment Group (N=53) | Standard Block Control Group (N=48)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) — Stomach distress or discomfort with a possible urge to vomit.
Seizure (Nervous system disorders) | 0 (0) | 1 (1) — A sudden burst of electrical activity in the brain possibly causing changes in behavior, movements, feelings and levels of consciousness

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-29): https://cdn.clinicaltrials.gov/large-docs/53/NCT05188053/Prot_SAP_000.pdf